CLINICAL TRIAL: NCT06559930
Title: Multiple Effects of Dual-Task Focused Training in Individuals with Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Yasemin Şahbaz, Dr. Lecturer, University of Beykent
Allocation: Not Applicable | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UBeykent-8
Record Dates: First submitted 2024-08-10; First posted 2024-08-19 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Chronic Stroke; Dual Task; Physiotherapy

STUDY DESIGN:
Intervention Model Description: Patients will be divided into 2 groups of 20 people each. The random division of the cases into groups and their treatments will be done by the same researchers. The evaluation will be carried out by another researcher to determine which groups will be divided into before and after the treatment. After the initial evaluations are made, a traditional recording program of 30 sessions will be applied to Group 1, every day for 6 weeks. The 2nd group is traditionally equalized and a dual-task-focused training program is applied twice a week for a total of 12 sessions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional Neurological Rehabilitation (Active Comparator): In-bed lower and upper extremity passive-active assisted-active ROM exercises Lower and upper extremity strengthening exercises with Theraband Electrotherapy will be applied to increase muscle strength in the tibialis anterior, quadriceps femoris, forearm extensors and elbow extensors.
  Interventions: Other: Traditional Neurological Rehabilitation
- Traditional Neurological Rehabilitation + Dual Task Focused Training (Experimental): In our Traditional Neurological Rehabilitation + Dual Task Focused Training group; Dual-task exercises were added in addition to the conventional treatment program.
  For dual task training:
  During in-bed exercises, the person will be asked to perform simple addition operations and rhythmic counting by 4 from 1 to 100.
  During balance and walking exercises, the person will be asked to count rhythmically by 2 from 1 to 40.
  Interventions: Other: Traditional Neurological Rehabilitation + Dual Task Focused Training

INTERVENTIONS:
Other: Traditional Neurological Rehabilitation + Dual Task Focused Training — Physiotherapy and rehabilitation after stroke increases joint movement, provides independence in activities of daily living, improves balance and coordination, manages pain, supports speech and swallowing skills, provides psychological support, and promotes social integration. Dual-task exercises, an important aspect of post-stroke rehabilitation, target both motor and cognitive functions. Dual tasks are activities that require performing two different tasks at the same time. These types of exercises are used to increase patients' attention, improve coordination, and help them perform daily living activities more effectively.
  Arms: Traditional Neurological Rehabilitation + Dual Task Focused Training
Other: Traditional Neurological Rehabilitation — Rehabilitation programs that start early after stroke and continue at regular intervals throughout life support the individual in regaining his quality of life and performing his daily functions. These programs can help patients increase their functional independence, improve their quality of life, and ensure their social integration. Physiotherapy and rehabilitation after stroke increases joint movement, provides independence in activities of daily living, improves balance and coordination, manages pain, supports speech and swallowing skills, provides psychological support, and promotes social integration.
  Arms: Traditional Neurological Rehabilitation

SUMMARY:
The aim of this study is to comprehensively investigate dual-task-focused training on balance, functionality, anxiety, healthy function and quality of life in chronic individuals. Stroke is a clinical condition that occurs as a result of deaths in the brain blood and is an important public health problem, ranking third among the causes of death in the world and first among the diseases that cause disability. There are a limited number of studies in the literature investigating the effectiveness of dual task training in stroke rehabilitation.

DETAILED DESCRIPTION:
Unlike other studies in the literature, this designed study evaluates balance, functionality, anxiety, cognitive functions and quality of life in addition to walking, making it unique. In the light of all this information, the hypothesis of the study is as follows: Application of dual-task-oriented training in addition to the regular physiotherapy program in individuals with chronic stroke affects balance, functionality, anxiety levels, cognitive functions and quality of life. It is planned to include 40 participants who meet the inclusion criteria in the study. After giving the necessary verbal and written information about the study, participants who receive informed consent will be randomized and divided into 2 groups of 20 people each. Group 1 will receive 30 sessions of traditional neurological rehabilitation program every day for 6 weeks. In Group 2, in addition to traditional neurological rehabilitation, a dual-task-oriented training program will be applied for a total of 12 sessions, twice a week. Participants will be evaluated twice, before and after treatment. Researchers will record personal information through a socio-demographic data form. Balance will be evaluated with the Berg Balance Test, functional status will be evaluated with the 10 Meter Walk Test and Timed Up and Go Test, anxiety level will be evaluated with the Beck Anxiety Scale, cognitive functions will be evaluated with the Verbal Fluency Test, and Standardized Mini Mental Test and quality of life will be evaluated with the Stroke Specific Quality of Life Scale.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to work
* Being between the ages of 40-70
* Being diagnosed with stroke
* Those who are not bedridden or wheelchair bound

Exclusion Criteria:

* People with sensory impairments (those with severe hearing and vision loss)
* Those with incompletely unioned fractures
* People with infection
* Those who have vestibular problems and balance problems
* Those who cannot cooperate due to psychiatric or cognitive problems
* Serious heart failure etc. those with systemic disease
* Bilateral involvement
* Accompanying serious orthopedic problem

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Berg Balance Test | 6 weeks
  The balance of the patients will be evaluated twice with the Berg Balance Test, before and after the treatment. Each item of the Berg Denf-ge Test, which consists of 4 items, is scored between 0-4. In this test, which measures a person's performance in different positions, higher scores indicate better balance. 56 points indicate no risk of falling, 41-56 points indicate a slight risk of falling, 21-40 points indicate a moderate risk of falling, and below 20 points indicate a high risk of falling. A Turkish validity and reliability study of the scale was conducted.
10 Meter Walking Test | 6 weeks
  The 10 meter walk test is a test generally used for physical capacity values. This test measures how long it takes an individual to travel a certain distance and can often be used in situations such as old age, detached parts, or certain health conditions. The application of the test is carried out by performing the following steps: Preparation of the test area, calculation of the starting position and walking speed.
Timed Up and Go Test Timed Up and Go Test Timed Up and Go Test | 6 weeks
  A chair and a stopwatch are required to perform the test, which evaluates fall risk and mobility in the elderly. The test is performed with the shoes the patient always uses and is told that he can use walking aids if he needs it. The 3-meter area in front of the chair is determined. The patient is asked to get up from the chair, walk this distance and sit down again. The elapsed time gives the result of the test. What to say to the patient: When I say start, do the following steps one by one; 1. Get up from the chair 2. Walk at your normal pace to the line ahead 3. Turn back 4. Walk at your normal pace towards the chair 5. Sit down. If an elderly individual completes this test in more than 12 seconds, there is a risk of falling.
Beck Anxiety Scale | 6 weeks
  Beck anxiety scale is a 4-point Likert type scale consisting of 21 questions that aims to measure the anxiety severity of the individual. Each question is scored between 0-3. A total score between 8 and 15 points from the scale indicates a low level of anxiety, a score between 16 and 25 indicates a moderate level of anxiety, and a score between 26 and 63 points indicates a high level of anxiety.
Verbal Fluency Test | 6 weeks
  It is a test frequently used in the evaluation of neurological disorders. In this test, people produce meaningful words from specified letters or specified categories (such as animal names, proper names, fruit) for a certain period of time. During our evaluation, people will be asked to count all the proper nouns that come to their mind for 1 minute. The test will be completed by scoring the number of words produced during this period, taking into account the number of words they count outside the category and the number of words they repeat.
Standardized Mini Mental Test | 6 weeks
  Standardized Mini Mental Test, a 30-item method, is a scale used to evaluate immediate memory, attention, recent memory and language functions. Due to its practicality and short-term applicability, it is widely used for screening purposes in samples thought to have cognitive impairment. The test has 5 subheadings. According to the scoring and evaluation method, orientation is grouped as 10 points, memory as 3 points, attention and calculation as 5 points, memory as 3 points, and language as 9 points. In general evaluation, 24-30 points indicate the normal value range, 18-23 points indicate a mild impact, and 0-17 points indicate a serious impact. As the total score increases, it indicates improvement.
Stroke-Specific Quality of Life Scale | 6 weeks
  The Stroke-Specific Quality of Life Scale (SSQOL) is used to assess quality of life. SSQOL consists of 12 subsections including energy, family roles, language, mobility, mood, personality, self-care, social roles, thinking, upper extremity function, vision and work-productivity, and a total of 49 questions. It is rated with a Likert type scoring from 1 to 5. The total score the patient can get is 49-245; As the score increases, it indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin ŞAHBAZ, Principal Investigator — Beykent University
Locations (1):
- Beykent University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayot M, Dujardin K, Tard C, Defebvre L, Bonnet CT, Allart E, Delval A. The interaction between cognition and motor control: A theoretical framework for dual-task interference effects on posture, gait initiation, gait and turning. Neurophysiol Clin. 2018 Dec;48(6):361-375. doi: 10.1016/j.neucli.2018.10.003. Epub 2018 Oct 26. PMID 30487064
- [Background] Plummer P, Iyigun G. Effects of Physical Exercise Interventions on Dual-Task Gait Speed Following Stroke: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2018 Dec;99(12):2548-2560. doi: 10.1016/j.apmr.2018.04.009. Epub 2018 May 5. PMID 29738743
- [Background] Meester D, Al-Yahya E, Dennis A, Collett J, Wade DT, Ovington M, Liu F, Meaney A, Cockburn J, Johansen-Berg H, Dawes H. A randomized controlled trial of a walking training with simultaneous cognitive demand (dual-task) in chronic stroke. Eur J Neurol. 2019 Mar;26(3):435-441. doi: 10.1111/ene.13833. Epub 2018 Nov 25. PMID 30308699
- [Background] Lee YS, Bae SH, Lee SH, Kim KY. Neurofeedback training improves the dual-task performance ability in stroke patients. Tohoku J Exp Med. 2015 May;236(1):81-8. doi: 10.1620/tjem.236.81. PMID 25985858
- [Background] Wong PL, Yang YR, Huang SF, Wang RY. Effects of Transcranial Direct Current Stimulation Followed by Treadmill Training on Dual-Task Walking and Cortical Activity in Chronic Stroke: A Double-Blinded Randomized Controlled Trial. J Rehabil Med. 2023 Mar 21;55:jrm00379. doi: 10.2340/jrm.v55.5258. PMID 36943024
- [Background] Green J, Forster A, Young J. Reliability of gait speed measured by a timed walking test in patients one year after stroke. Clin Rehabil. 2002 May;16(3):306-14. doi: 10.1191/0269215502cr495oa. PMID 12017517
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Hong SY, Moon Y, Choi JD. Effects of Cognitive Task Training on Dynamic Balance and Gait of Patients with Stroke: A Preliminary Randomized Controlled Study. Med Sci Monit Basic Res. 2020 Aug 10;26:e925264. doi: 10.12659/MSMBR.925264. PMID 32773732